CLINICAL TRIAL: NCT05708300
Title: Novel Insight in pathologiCal and clinicAl Attributes in Response to mepoLizumab Treatment in Patients With Chronic rhInosinusitis With Nasal pOlyPs With or Without bronchIal Asthma on a Long-term Basis (CALIOPI STUDY)
Brief Title: Biomarkers of Response to Mepolizumab Treatment in Patients With Nasal Polyps With or Without Bronchial Asthma
Acronym: CALIOPI
Status: Recruiting | Type: Observational
Sponsor: Aristotle University Of Thessaloniki (Other)
Collaborators: Department of Otorhinolaryngology, Head and Neck Surgery, George Papanikolaou Hospital (Unknown); Department of Otorhinolaryngology, Democritus University of Thrace, Alexandroupolis (Unknown); Department of Pulmonology, Democritus University of Thrace, Alexandroupolis (Unknown); Respiratory Medicine Department, University of Ioannina, Faculty of Medicine (Unknown); Department of Respiratory Medicine, National and Kapodistrian University of Athens (Unknown); Department of Allergy and Clinical Immunology, 424 General Military Training Hospital (Unknown); Department of Otolaryngology, Head and Neck Surgery, Sotiria General Hospital (Unknown); Pulmonary and Respiratory Failure Department, National and Kapodistrian University of Athens (Unknown)
Responsible Party: Principal Investigator, Associate Prof Konstantinos Porpodis, Associate Professor of Pulmonology, Aristotle University Of Thessaloniki
Other Study IDs: Study 14879
Record Dates: First submitted 2022-12-29; First posted 2023-02-01 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Chronic Rhinosinusitis With Nasal Polyps; Asthma
Keywords: Chronic Rhinosinusitis; Nasal Polyps; Asthma
MeSH Terms: conditions — Asthma; Nasal Polyps | interventions — mepolizumab; Biological Products; Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — blood,
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- chronic rhinosinusitis with nasal polyps with bronchial asthma: Patients with chronic rhinosinusitis with nasal polyps with bronchial asthma will be administered Mepolizumab (100 MG), subcutaneusly every 30 days
  Interventions: Drug: Mepolizumab 100 MG [Nucala]
- chronic rhinosinusitis with nasal polyps without bronchial asthma: Patients with chronic rhinosinusitis with nasal polyps without bronchial asthma will be administered Mepolizumab (100 MG), subcutaneusly every 30 days
  Interventions: Drug: Mepolizumab 100 MG [Nucala]

INTERVENTIONS:
Drug: Mepolizumab 100 MG [Nucala] — subcutaneous injection once a month
  Other Names: biologicals/vaccine

SUMMARY:
Mepolizumab is a biologic agent already approved for severe asthma. Recently, there is increasing evidence concerning the benefit of anti-IL5 treatments upon patients with nasal polyposis with or without severe asthma.

The novelty of this project is that no biologic agent has yet been fully investigated to identify any biomarkers of response for patients with nasal polyps with or without asthma including sinonasal tissue remodeling a key element in the resultant histopathological changes of the inflammation. The investigation of airway remodeling of various locations (nose and bronchus) under mepolizumab treatment will be our primary objective on the long-term basis of 156 weeks of treatment.

Endobronchial and nasal biopsies will be performed as routine care for tissue evauation and disease investigation for every patient.

Besides, the united airways will provide better guidance for medical treatment of chronic rhinosinusitis (CRS) patients with nasal polyps (CRSwNP) and asthma.

The initial idea is based on investigating the characteristics that could predict the effectiveness of mepolizumab on patients with nasal polyposis with or without asthma. Patients will receive 39 doses of mepolizumab for 156 weeks. An additional aim of this study is to identify characteristics of non-responders and responders to mepolizumab. Responders will be identified based on airway remodeling status, biomarkers in tissue and secretion samples and on the reduction of the need of surgery through Lund-Kennedy endoscopic score, Lund-Mackay score and patient's clinical status in the 6th, 12th and 36th month after the initiation of treatment.

Regarding the unified airway system, nose and pharyngeal microbiome will be evaluated before and after 52 weeks of mepolizumab treatment in patients with nasal polyps whereas in patients with nasal polyps and asthma bronchus microbiome will also be evaluated. Lung samples will help gain information about the inflammatory profile and local microbiome of CRSwNP patients with asthma through molecular and cellular assays. The human Pharyngeal Microbiome might play a protective role in Respiratory Tract Infections and it has been reported that the microbiome provides critical signals to promote maturation of immune cells and differentiation of the tissue. Thus, we will make an effort to correlate microbiome of various locations with clinical and laboratory characteristics of responders and non-responders to mepolizumab treatment.

DETAILED DESCRIPTION:
Hypothesis Identification of pathological and clinical characteristics of responders and non-responders to mepolizumab treatment in patients with chronic rhinosinusitis with nasal polyps with or without bronchial asthma regarding the airway remodeling, inflammatory cells and other biomarkers on a long-term basis.

Objectives/Endpoints

The primary objectives of this study are:

1. Evaluation of the airway remodeling in various anatomic locations of the airways (nose, bronchus) at baseline-before treatment initiation and after 156 weeks of mepolizumab treatment.
2. Identification of any characteristics in microbiome of various locations (nose, pharyngeal, bronchus) in responders and non-responders to mepolizumab treatment.

The key secondary objectives of this study are:

1. Combination of selected inflammatory biomarkers of various anatomic locations in the airways in tissue and secretion samples to identify non-responders and responders to mepolizumab after 152 weeks of mepolizumab treatment.
2. To demonstrate the effect of mepolizumab treatment in patients with nasal polyps with or without bronchial asthma through the reduction of patients requiring surgery after 52 weeks of treatment taking into consideration the airway remodeling, inflammatory cells and biomarkers of inflammation and clinical characteristics.

   Other objectives/endpoints Any improvement in respiratory parameters in asthma control and in patients' quality of life including sleep quality during mepolizumab treatment in patients with nasal polyps with or without bronchial asthma.

   Any possible biomarkers of response considering nasal polyps and bronchial asthma as a unified airway disease after 52 weeks of treatment and after 156 weeks of treatment.

   Characterization of patients' compliance to mepolizumab doses for 156 weeks.

   Study design and Methods A phase IV study, where patients will be collected from outpatient clinics of Bronchial Asthma and of Ear Nose Throat from each site which cover the population of Greece. Due to the unknown situation concerning Covid-19 pandemic, we assume that this clinical study does not interfere with the workload in our Clinics.

   Overall, this is a prospective multicenter study including 7clinics. The study will include a screening period of up to 2 weeks to assess eligibility and obtain written informed consent and a mepolizumab treatment period of 156 weeks.

   Sampling method, number of subjects and timelines Study population The study population will consist of approximately 57 patients with nasal polyposis with or without bronchial asthma receiving mepolizumab for three years aged 18 and above (no children). Clinical evaluation of patients with nasal polyposis with or without asthma will be made according to the European Position Paper on Rhinosinusitis and Nasal Polyps. Besides, standard of care for our patients apart from mepolizumab may include ICS, anti-histamine or LTRAs.

   Target enrolment Our target sample size was calculated on the basis that 57 patients was the minimum sample size, computed for reticular basement membrane thickness from g-power analysis (as described in the paragraph of calculation of sample size). We add an additional 5% to ensure the validity of the results in case of potential patient withdrawals during our perspective study.

   Study participation, assessment and follow up:

   Vital signs, will be performed at site visits at screening visit, at baseline and every 3 months. Measurements will include systolic and diastolic blood pressure, pulse rate and body temperature.

   Height in centimeters (cm) and body weight in kilograms (kg) will be measured at screening visits. Body Mass Index (BMI) will be calculated as the weight in kg divided by the height in meters squared

   Laboratory evaluation (Hematology, Blood chemistry, Urinalysis) includes venous blood and urine will be collected at baseline. Collection of urine for female subjects will also evaluate pregnancy. IgE levels will be evaluated at screening visit using immunoCAP tests and will be reported as IU/mL.

   Questionnaires The following will be administered: 1) the Asthma Control Questionnaire (ACQ-5) and Asthma Control Test (ACT) to assess current asthma control; 2) the Asthma Quality of Life Questionnaire (AQLQ+12) to assess quality of life and psychological morbidity. To further asses sleeping quality 1) Athens Insomnia Scale (AIS), 2) Epworth Sleepiness Scale (ESS), 3) St. George's Respiratory Questionnaire (SGRQ) and 4) WHO (Five) Well-Being Index (WHO-5), 5) Fatigue Severity Scale (FSS), 6) Visual Analogue Scale (VAS) score, 7) SinoNasal Outcome Test (SNOT-22) score, 8) University of Pennsylvania Smell Identification Test (UPSIT) score.

   FeNO Exhaled nitric oxide (NO) will be measured at baseline and every 6 months according to the American Thoracic Society Guidelines and as specified by the manufacturer. FeNO levels will be reported as parts per billion. Measurements will be made before spirometry is performed.

   Blood eosinophil levels Venous blood samples will be retrieved between 8 to 10 am, at baseline and every 3 months during the 156-week period with mepolizumab treatment. Absolute blood eosinophil count will be reported as cells/μl.

   Spirometry Spirometry will be conducted, using the site's own equipment at the visits (baseline and every 3 months) as specified in the table 1. All clinic visits must occur in the morning. During the treatment period the spirometry will meet the current ATS/ERS guidelines and the spirometer must produce a printout of all data generated, which should be stored in the subject's notes. The spirometer will be calibrated in accordance with the manufacturer's instructions. Spirometry must be performed at the same time (±1 hour) of the Visit 0 spirometry. Subjects should try to withhold short-acting beta-2-agonists (SABAs) for ≥4 hours and LABAs for ≥15 hours prior to clinic visit, if possible (GINA 2019). Assessments to be recorded will include FEV1, FVC, FEV1/FVC%, PEF and FEF25-75. Post-bronchodilator measurements will be taken at every visit, using 200-400mcg albuterol or equivalent.

   Impulse Oscillometry Impulse Oscillometry (IOS) will be conducted at baseline, after 52 weeks of treatment and after 156 weeks of treatment.

   Lund Mackay Score Lund-Mackay computed tomography (CT) score will be evaluated by CT sinus at baseline, after 52 and 156 weeks of treatment as specified in table 1. Preoperative and follow up CT sinus are used in clinical practice in CRS patients as standard of care in sponsor's country (radiation dose about 50mGy). Lund-Mackay CT staging will be evaluated blindly by 2 different clinicians.

   Peak nasal inspiratory flow (PNIF) PNIF will be applied at baseline and every 6 months until 156-week of treatment. PNIF will be evaluated using Olympus ENF type P4 fibroscope and a Clement Clark International Limited model IN-CHECK ORAL ATM device.

   Anterior Rhinomanometry Anterior Rhinomanometry will be conducted at baseline and every 6 months until 156-week of treatment by rhinomanometry system PDD-301/sr.

   Therapy with biologics Upon completion of the screening visits the participant may initiate treatment with biologic therapy (mepolizumab) within a month. During therapy subjects will be under the care of the pulmonologist who had referred them to the research group for taking part into the study. These pulmonologists will be termed as 'associate pulmonologists. Treatment will be provided as per product manufacturer instructions.

   Associate pulmonologists and otorhinologists providing biologic treatment during the study will require to sign an agreement to conduct the study in compliance with the protocol, to acknowledge that he/she is responsible for medical conduct and for study conduct, and to ensure that the associate (and their colleagues and employees) assisting in the conduct of the study are informed about their obligations.

   Mechanisms will be in place to ensure that associate staff receives the appropriate information and support by the research group throughout the study.

   Follow up during biologic therapy: At initiation and at every visit for biologic therapy administration collection of information (see table 1) will be performed by the associate pulmonologist, and with support by the research group if requested by the associate pulmonologist e.g., researchers via telephone or face-to-face contact will interview the patient. Furthermore, compliance will be recorded form the physician based on patient's oral confirmation. Date form of drug administration will be recorded at every visit, as well as immediate and delayed adverse effects.

   Safety monitoring Recorded adverse events (AEs) will be monitored and collated as required in study reports.

   Adverse events An adverse event is the appearance or worsening of any undesirable sign, symptom, or medical condition occurring after starting the study entry. Medical conditions/diseases present before starting study drug are only considered adverse events if they worsen after starting study drug. Abnormal laboratory values or test results constitute adverse events only if they induce clinical signs or symptoms, are considered clinically significant, or require therapy. Also, adverse events related to Covid-19 are included. If a partner pulmonologist or research staff becomes aware of an AE associated with a product, it can be reported to the manufacturer according to their local standard practice for spontaneous AE reporting. A copy of the report should also be sent to the study coordinator. Serious adverse events (SAE) will be reported in the eCRF pages and within 24 hours all the investigators will have the responsibility to inform the Central Committee in Thessaloniki. Then the Central Committee will inform the scientific board and the Greek Medical Agency. Also, medical and scientific judgment will be exercised by the principal investigator of each center with the Central Committee, in deciding whether the subject should stop the treatment or not.

   Independent Data Monitoring Committee/Data and Safety Monitoring Board (IDMC/ DSMB) is the central research personnel in Thessaloniki (Central Committee). For a successful monitoring of protocol assessments, IDMC/DSMB will schedule a phone-call every month to all the sites included.

   Konstantinos Porpodis -Principal Investigator (Associate Professor, Pulmonary Department, Aristotle University of Thessaloniki, George Papanikolaou Hospital, Thessaloniki), Kalliopi Domvri - Clinical Research Associate-Study Manager-Sub Investigator, Laboratory of Histology-Embryology, Medical School, Aristotle University of Thessaloniki.

   Pregnancy report Initially, female patients at screening will have to do a pregnancy test. During treatment, if a female subject reports a pregnancy to us, she will be asked to withdraw from the study (to prevent bias) Then, she will be asked if she would like to keep getting the treatment outside of this protocol and be monitored at each center's outpatient clinic.

   Pre-screening and Screening Failures Subjects will be assigned a study number at the time of signing the consent. Subjects who signed but do not progress to the screening visits assessment will be deemed a pre-screen failure. No data will be captured in the database for these subjects.

   Subjects that complete at least one of the two screening visits, but do not initiate biologic therapy will be designated as screening failures.

   Information to be collected for pre-screening and screening failures will be detailed in the database completion.

   Withdrawal Visit If a participant decides to withdraw from the study during follow-up (for any reason other than loss to follow up), they may be asked to attend a withdrawal visit (if deemed necessary by investigator and subject to consent). During the visit, the participant may be asked questions about their current conditions as part of clinical information collection such as: asthma and nasal symptoms, exacerbations and the progression of treatment being received.

   Blood samples' collection and processing Blood samples will be collected at baseline visit, at 6 months and after treatment completion.

   Induced sputum Induced sputum will be performed at baseline before treatment initiation and after 52 and 156 weeks of treatment according to the ERS Task Force report where a detailed expert consensus-based recommendation for induced sputum processing is suggested. After collecting the induced sputum, the supernatant of the sample will be stored at -20° C in eppendorf tubes till the analysis was done.

   Bronchoscopy, bronchial/nasal biopsies and washing samples' collection and processing Endoscopy with bronchial biopsies, bronchial washing sample will be performed upon patient's written consent. In specific, a separate inform consent will be included to be signed from each patient. Bronchoscopy will be performed at three time-points (baseline before treatment initiation, after 52 weeks of treatment and after 156 weeks of treatment). Flexible bronchoscopy and diagnostic techniques were performed under monitored anesthesia care as recommended by the American Thoracic Society and the British Thoracic Society.

   Nasal biopsies will be performed at baseline visit, after 52 and 156 weeks of treatment upon patient's written consent. Endoscopic surgical procedure will be performed with nasal scissors by cutting the tissue and then removing the sample. The method will be performed as a Functional endoscopic sinus surgery (FESS), a minimally invasive technique under direct visualization. The endoscopic procedure requires local anesthetic. The specific features that will be identified and assessed during the examination are the middle turbinate and the middle meatus (osteomeatal complex), anatomic obstruction, mucopus and nasal polyps.

   After the endoscopic procedures, tissue samples will be fixed in inflation or immersion using formaldehyde or glutaraldehyde and embedded in paraffin. Airways will be systematically sampled or obtained during diagnostic dissection at the discretion of the pathologist. Airway remodeling will be evaluated not only by optical microscopy but also by electron microscopy.

   Finally, bronchial washing samples will be immediately transported to the laboratory, to be stored at -80 degrees. Examination of bronchial washing fluids will be performed at a later stage to determine several biomarkers by RT-PCR, ELISA and flow cytometry as described in the next paragraph.

   For the evaluation of biomarkers of inflammation in tissue, blood and other biological fluids, Flow Cytometry Analysis (FACS) with beads or ELIZA method will be performed. Immunophenotype will be analyzed by FACS. Expression of biomarkers will be evaluated by RT-PCR. Biomarker will be evaluated before the initiation, after 1-year and after 156-week of mepolizumab treatment.

   Microbiome analysis Microbiome samples will be taken at baseline and after 52-weeks of treatment. Quantification of total bacteria, specific taxa and butyrate production capacity will be carried out by qPCR using a BioRad iCycler iQ thermal cycler system (BioRad, Hercules, CA).

   Allergy testing (If applicable) The patients' atopic status will be evaluated (if not available) at screening visit by the skin prick test (SPT) to a standard panel of aeroallergens for detecting total IgE antibodies against various common inhalant allergens.

   Sample size calculation G power analysis Sample size is calculated using the G*Power software (Die Heinrich-Heine-Universität Düsseldorf, Germany). The difference in reticular basement membrane thickness before and after mepolizumab treatment for the investigation of airway remodeling in patients with chronic rhinosinusitis with nasal polyps with or without bronchial asthma is one of our primary endpoints. In the study by Diver et al, it has been reported that reticular basement membrane thickness before and after tezepelumab treatment was found 3.86 ± 1.54 vs 3.35 ± 1.34 respectively. Using this data and a two-sided test, with a power at 0.95 and a level of statistical significance at 0.05, we calculated an effect size of 0.49, which indicated a total sample size of 57 participants.

   Sarah Diver, Latifa Khalfaoui, Claire Emson, Sally E Wenzel, Andrew Menzies-Gow, Michael E Wechsler, James Johnston, Nestor Molfino, Jane R Parnes, Ayman Megally, Gene Colice, Christopher E Brightling, CASCADE study investigators. Effect of tezepelumab on airway inflammatory cells, remodelling, and hyperresponsiveness in patients with moderate-to-severe uncontrolled asthma (CASCADE): a double-blind, randomised, placebo-controlled, phase 2 trial. Lancet Respir Med. 2021 Nov;9(11):1299-1312.

   Statistical Plan Analysis Statistical analysis will be performed using the SPSS (version 21.0 IBM SPSS statistical software, Armonk, NY, USA). Categorical variables will be stated as numbers (n) and percentages (%), continuous variables as mean ± SD if normally distributed, or median and interquartile ranges if otherwise. Where necessary variables without a normal distribution will be transformed. P < 0.05 was accepted as statistically significant. Shapiro-Wilk test will be performed in order to separate parametric from non-parametric variables. Paired-Samples T Test for parametric or Wilcoxon Signed Ranks test for non-parametric variables will be used to detect differences in the variables measured before and after Mepolizumab treatment in CRS patients with nasal polyps with or without asthma in both histopathological, blood or clinical parameters.

   There is no comparator arm as every patient is control to himself. There are baseline characteristics (clinical and laboratory biomarkers) that are going to be measured at baseline, every 6 months, after 52 and 156 weeks of treatment completion. Primary end-point is changes in the airway remodeling both in nose and bronchus.

   Study endpoints also include the analysis of all those biomarkers as the identification of the characteristics of non-responders and super-responders. Also, secondary endpoints include the evaluation of the biomarkers mentioned in the methods as assessments. Statistical analysis will be performed initially with the number of patients that have completed the 52-week period of treatment and the 156-week. Secondly, patients that have not completed the treatment will be analyzed separately and finally these two groups are going to be compared to each other.

   Airway remodeling and overall response to treatment and in one and three years (from baseline to 1-year post treatment initiation) for each outcome will be measured with paired test of dependent samples (parametric and non-parametric paired tests) in each patient. Then response to treatment will be defined as the change (absolute and % change) of the outcome in one and three years. We will assess predictors influencing response to treatment (change) such as biomarkers by using multiple regression models for each clinicopathological outcome. For outcomes with more than 2 observations per subject during the study period we will use mixed models using the repeated measurements of the outcome. All tests will be 2-sided with a statistical significance level at 5%.

   Database

   Data collection method:

   An electronic data collection platform will be the method used at baseline every 3 months until 1 year follow up for this database. During treatment visits paper forms/questionnaires will be completed by the associate pulmonologist/otorhinolaryngologist. Each site will entry specific data in an electronic database. Each patient is uniquely identified by a Subject number which is composed by the site number assigned by the responsible monitoring site and a sequential number assigned by the investigator. Upon signing the informed consent form, the patient is assigned the next sequential number by the investigator. The site must contact the central research personnel and provide the requested identifying information for the patient as registered into the electronic database. The treatment visit forms will also be sent to the central research personnel. The authorized study personnel will be responsible for data collection, editing, and also protecting the data being collected at their own site and the database is backed up on a daily basis. Quality review/control will be the joint responsibility of all individuals involved and the central research personnel [data custodian].

ELIGIBILITY:
Inclusion Criteria:

* Adult patients > 18 years with bilateral Nasal Polyps
* Symptoms VAS scores (for nasal obstruction, hyposmia, post-nasal drip, sneezing, rhinorrhea; 0-10 for each symptom) > 24 in spite of treatment with standard of care treatment.
* Patients with bilateral sinonasal polyps with a need for surgery as described by: Lund-Mackay score > 4, Lund Kennedy score > 6, a minimum total Nasal polyp score of 5 out of a maximum score of 8 at screening, ongoing symptoms for at least 12 weeks prior to screening,
* Concerning patients with asthmatics with nasal polyps: subjects must have a medical history of asthma as confirmed by asthma related symptoms and by bronchodilator response (BDR) (GINA 2022) or positive methacholine challenge according to ERS guidelines.

Exclusion Criteria:

* Pregnant or nursing women, or women of child-bearing potential.
* Biologic therapy (eg: Omalizumab, Mepolizumab, Reslizumab, Dupilumab) or previous treatment with Mepolizumab
* Allergen immunotherapy in the past 6 months
* Systemic corticosteroid treatment for other chronic conditions (i.e.: autoimmune disorders, tumors, etc)
* Prior/concomitant therapy: use of immunosuppressive medication (including but not limited to: methotrexate, troleandomycin, cyclosporine, azathioprine, or any experimental anti-inflammatory therapy) within 3 months prior to Visit 1 and during the study period.
* Evidence of active systemic immunodepression (i.e..: primary or secondary immunodeficiency)
* History of malignancy of any organ system or any other serious co-morbidities defined by the treating physician.
* Primary diagnosis of lung disease other than asthma (chronic obstructive lung disease (COPD), asthma-COPD overlap (ACO), interstitial lung disease, sarcoidosis, bronchiectasis, cystic fibrosis, primary ciliary dyskinesia, active tuberculosis, allergic bronchopulmonary aspergillosis (ABPA), current lung cancer or other blood, lymphatic or solid organ malignancy, autoimmune diseases of the skin, muscle-skeletal or gastrointestinal system needing systemic corticosteroids, immunosuppressants or biologic treatment as well as individuals with granulomatosis with polyangiitis (Wegener's granulomatosis) and eosinophilic granulomatosis polyangiitis (Churg-Strauss syndrome).
* Nasal polyps' or Asthma exacerbation, within 12 weeks prior to screening that required oral corticosteroids over 3 days or hospitalization or emergency room visit.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Study population The study population will consist of approximately 57 patients with nasal polyposis with or without bronchial asthma receiving mepolizumab for a year aged 18 and above (no children). Clinical evaluation of patients with nasal polyposis with or without asthma will be made according to the European Position Paper on Rhinosinusitis and Nasal Polyps. Besides, standard of care for our patients apart from mepolizumab may include ICS, anti-histamine or LTRAs.
Sampling Method: Non-Probability Sample
Enrollment: 57 (Estimated)
Dates: Start 2024-02-23 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in Basement Membrane Thickness | through study completion, 156 weeks
  The identification of clinical characteristics of non-responders and super-responders.
  Anwers whether change basement membrane thickness can predict therapeutic response of mepolizumab among patients.
Change in smooth muscle cell mass | through study completion, 156 weeks
  The identification of clinical characteristics of non-responders and super-responders.
  Anwers whether change in smooth muscle cell mass can predict therapeutic response of mepolizumab among patients.
Change in microbiome | through study completion, 156 weeks
  Answers whether there is a microbiome signature at baseline that can predict therapeutic response of mepolizumab among patients.
  The identification of clinical characteristics of non-responders and super-responders.

SECONDARY OUTCOMES:
Change of cytokine and protein levels in serum | through study completion, 156 weeks
  To identify any possible biomarkers of response of non-responders versus super-responders.
Change in exacerbation rate | through study completion, 156 weeks
  Mesurement of the change in exacerbation rate in patients with nasal polyps with asthma under mepolizumab treatment for 156 weeks of treatment
Change in requiring surgery | through study completion, 156 weeks
  Mesurement of the requirement of surgery in patients with nasal polyps with or without asthma under mepolizumab treatment for 156 weeks of treatment
Change of cytokine and protein levels in bronchial washing | through study completion, 156 weeks
  To identify any possible biomarkers of response of non-responders versus super-responders.

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos Porpodis, Assoc Prof, Principal Investigator — Pulmonary Clinic, Aristotle University of Thessaloniki, George Papanikolaou Hospital
Locations (2):
- Greece (2):
  - Pulmonary Clinic of Aristotle University of Thessaloniki, George Papanikolaou Hospital, Thessaloniki, Exochi
  - University Pulmonary Clinic, George Papanikolaou Hospital, Thessaloniki

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Fokkens WJ, Lund VJ, Hopkins C, Hellings PW, Kern R, Reitsma S, Toppila-Salmi S, Bernal-Sprekelsen M, Mullol J, Alobid I, Terezinha Anselmo-Lima W, Bachert C, Baroody F, von Buchwald C, Cervin A, Cohen N, Constantinidis J, De Gabory L, Desrosiers M, Diamant Z, Douglas RG, Gevaert PH, Hafner A, Harvey RJ, Joos GF, Kalogjera L, Knill A, Kocks JH, Landis BN, Limpens J, Lebeer S, Lourenco O, Meco C, Matricardi PM, O'Mahony L, Philpott CM, Ryan D, Schlosser R, Senior B, Smith TL, Teeling T, Tomazic PV, Wang DY, Wang D, Zhang L, Agius AM, Ahlstrom-Emanuelsson C, Alabri R, Albu S, Alhabash S, Aleksic A, Aloulah M, Al-Qudah M, Alsaleh S, Baban MA, Baudoin T, Balvers T, Battaglia P, Bedoya JD, Beule A, Bofares KM, Braverman I, Brozek-Madry E, Richard B, Callejas C, Carrie S, Caulley L, Chussi D, de Corso E, Coste A, El Hadi U, Elfarouk A, Eloy PH, Farrokhi S, Felisati G, Ferrari MD, Fishchuk R, Grayson W, Goncalves PM, Grdinic B, Grgic V, Hamizan AW, Heinichen JV, Husain S, Ping TI, Ivaska J, Jakimovska F, Jovancevic L, Kakande E, Kamel R, Karpischenko S, Kariyawasam HH, Kawauchi H, Kjeldsen A, Klimek L, Krzeski A, Kopacheva Barsova G, Kim SW, Lal D, Letort JJ, Lopatin A, Mahdjoubi A, Mesbahi A, Netkovski J, Nyenbue Tshipukane D, Obando-Valverde A, Okano M, Onerci M, Ong YK, Orlandi R, Otori N, Ouennoughy K, Ozkan M, Peric A, Plzak J, Prokopakis E, Prepageran N, Psaltis A, Pugin B, Raftopulos M, Rombaux P, Riechelmann H, Sahtout S, Sarafoleanu CC, Searyoh K, Rhee CS, Shi J, Shkoukani M, Shukuryan AK, Sicak M, Smyth D, Sindvongs K, Soklic Kosak T, Stjarne P, Sutikno B, Steinsvag S, Tantilipikorn P, Thanaviratananich S, Tran T, Urbancic J, Valiulius A, Vasquez de Aparicio C, Vicheva D, Virkkula PM, Vicente G, Voegels R, Wagenmann MM, Wardani RS, Welge-Lussen A, Witterick I, Wright E, Zabolotniy D, Zsolt B, Zwetsloot CP. European Position Paper on Rhinosinusitis and Nasal Polyps 2020. Rhinology. 2020 Feb 20;58(Suppl S29):1-464. doi: 10.4193/Rhin20.600. PMID 32077450
- [Result] Albers FC, Papi A, Taille C, Bratton DJ, Bradford ES, Yancey SW, Kwon N. Mepolizumab reduces exacerbations in patients with severe eosinophilic asthma, irrespective of body weight/body mass index: meta-analysis of MENSA and MUSCA. Respir Res. 2019 Jul 30;20(1):169. doi: 10.1186/s12931-019-1134-7. PMID 31362741
- [Result] Postma DS, Brightling C, Baldi S, Van den Berge M, Fabbri LM, Gagnatelli A, Papi A, Van der Molen T, Rabe KF, Siddiqui S, Singh D, Nicolini G, Kraft M; ATLANTIS study group. Exploring the relevance and extent of small airways dysfunction in asthma (ATLANTIS): baseline data from a prospective cohort study. Lancet Respir Med. 2019 May;7(5):402-416. doi: 10.1016/S2213-2600(19)30049-9. Epub 2019 Mar 12. PMID 30876830
- [Result] Detoraki A, Tremante E, D'Amato M, Calabrese C, Casella C, Maniscalco M, Poto R, Brancaccio R, Boccia M, Martino M, Imperatore C, Spadaro G. Mepolizumab improves sino-nasal symptoms and asthma control in severe eosinophilic asthma patients with chronic rhinosinusitis and nasal polyps: a 12-month real-life study. Ther Adv Respir Dis. 2021 Jan-Dec;15:17534666211009398. doi: 10.1177/17534666211009398. PMID 33910399
- [Result] Kuo CW, Liao XM, Huang YC, Chang HY, Shieh CC. Bronchoscopy-guided bronchial epithelium sampling as a tool for selecting the optimal biologic treatment in a patient with severe asthma: a case report. Allergy Asthma Clin Immunol. 2019 Nov 27;15:76. doi: 10.1186/s13223-019-0378-6. eCollection 2019. PMID 31798645
- [Result] Donnell NJ, Marino MJ, Zarka MA, Lal D. Histopathological characteristics of surgical tissue from primary vs recurrent chronic rhinosinusitis with nasal polyposis patients. Laryngoscope Investig Otolaryngol. 2020 Feb 7;5(1):5-10. doi: 10.1002/lio2.358. eCollection 2020 Feb. PMID 32128424
- [Result] Diver S, Khalfaoui L, Emson C, Wenzel SE, Menzies-Gow A, Wechsler ME, Johnston J, Molfino N, Parnes JR, Megally A, Colice G, Brightling CE; CASCADE study investigators. Effect of tezepelumab on airway inflammatory cells, remodelling, and hyperresponsiveness in patients with moderate-to-severe uncontrolled asthma (CASCADE): a double-blind, randomised, placebo-controlled, phase 2 trial. Lancet Respir Med. 2021 Nov;9(11):1299-1312. doi: 10.1016/S2213-2600(21)00226-5. Epub 2021 Jul 10. PMID 34256031